CLINICAL TRIAL: NCT04251780
Title: Changes in Tissue Potassium Amount Before and After Treatment of Primary Hyperaldosteronism Assessed by 39K-MRI
Brief Title: Tissue K+ in Primary Hyperaldosteronism
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: ConnK+
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Primary Hyperaldosteronism; Electrolyte Disturbance
Keywords: Hyperaldosteronism; Potassium; Magnetic Resonance Imaging
MeSH Terms: conditions — Hyperaldosteronism | interventions — Adrenalectomy; Dosage Forms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples Without DNA — Urine and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Primary Aldosteronism: Patients with primary Aldosteronism will either be treated by adrenalectomy (in case of unilateral adrenal disease) or receive medical treatment (Spironolactone/Eplerenone; bilateral hyperplasia) as specified in the endocrinological guideline (J Clin Endocrinology & Metabolism, May 2016). Before and after intervention tissue sodium and tissue potassium amount will be assessed by MRI.
  Interventions: Procedure: Surgical Treatment of Primary Aldosteronism; Drug: Drug treatment of Primary Aldosteronism
- Control group: Healthy participants, age- and gender-matched with the Primary Aldosteronism patients. Tissue sodium and tissue potassium amount of the healthy control group will be assessed by MRI and compared to the tissue sodium and potassium amount of the patients with Primary Aldosteronism before treatment.

INTERVENTIONS:
Procedure: Surgical Treatment of Primary Aldosteronism — Surgery of an unilateral adrenal disease
  Other Names: Adrenalectomy
  Groups: Patients with Primary Aldosteronism
Drug: Drug treatment of Primary Aldosteronism — Treatment of Primary Aldosteronism with Spironolactone or Eplerenone.
  Other Names: Medication
  Groups: Patients with Primary Aldosteronism

SUMMARY:
Recent human studies found tissue sodium storage in patients with hyperaldosteronism that could be detected non-invasively by 23Na-MRI. Tissue sodium accumulation could be mobilized upon treatment of hyperaldosteronism. Besides, former animal studies applying chemical electrolyte analysis indicate that this aldosterone induced sodium storage might be accompanied by intracellular potassium loss. Wether such an intracellular tissue potassium loss occurs in vivo in patients with hyperaldosteronism and if this deficiency can be corrected by treatment is unclear. The investigators will employ 39K-MR Imaging at 7Tesla to further assess this hypothesis.

DETAILED DESCRIPTION:
Patients diagnosed with primary hyperaldosteronism (PA) will be prospetively investigated using 23Na-MRI and 39K-MRI at 7 Tesla to assess tissue sodium and potassium content (prospective observational study). Measurements will be conducted before treatment of hyperaldosteronism and three to four months after adrenal surgery or medical treatment (Spironolactone or Eplerenone). Furthermore, blood pressure, body water distribution (by bioimpedance spectroscopy), pulse wave velocity and serum electrolytes will be assessed.

Additionally, we will conduct a case-control study and compare PA patients before treatment with age- and gender matched healthy control participants. In this study group 23Na-MRI and 39K-MRI at 7 Tesla will be conducted to assess tissue sodium and potassium content using the same MRI protocols as in PA patients. Blood pressure, body water distribution (by bioimpedance spectroscopy), pulse wave velocity and serum electrolytes will be also examined.

ELIGIBILITY:
Inclusion Criteria for patients with Primary Aldosteronism:

* Primary Aldosteronism diagnosed according to the endocrinological guideline (J Clin Endocrinology & Metabolism, May 2016) without specific medication
* Age > 18 years

Exclusion Criteria for patients with Primary Aldosteronism:

* Chronic kidney disease ≤ 3b (estimated GFR <45 ml/min according to CKD-EPI)
* Active malignancy
* Severe congestive heart failure (NYHA III and IV)
* Liver cirrhosis (Child B and C)
* Acute infection
* Recent major surgical procedures (<3 months)
* Pregnancy
* Contraindications for MRI measurements: cardiac pacemaker, claustrophobia, etc.

Inclusion Criteria for healthy control participants:

- Age > 18 years

Exclusion Criteria for healthy control participants:

* Medical history of chronic disease (such as diabetes, hypertension, chronic kidney disease etc.)
* regular medication
* blood pressure ≥ 140/90 mmHg
* Pregnancy
* Contraindications for MRI measurements: cardiac Pacemaker, claustrophobia, etc.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Primary Aldosteronism Healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Tissue potassium content | 3-6 months after intervention
  1. Change in tissue potassium content measured by MRI before and after treatment of Primary Aldosteronism
  2. Difference in tissue potassium content between patients with Primary Aldosteronism before treatment and healthy control subjects

SECONDARY OUTCOMES:
Tissue sodium content | 3-6 months after intervention
  1. Change in tissue sodium content measured by MRI before and after treatment of Primary Aldosteronism
  2. Difference in tissue sodium content between patients with Primary Aldosteronism before treatment and healthy control subjects
Blood pressure | 3-6 months after intervention
  Change in blood pressure (systolic/diastolic/mean) before and after treatment of Primary Aldosteronism
Water balance | 3 - 6 months after intervention
  1. Change in water distribution (intra-/extracellular water, total water, overhydration) assessed by bioimpedance spectroscopy before and after treatment of Primary Aldosteronism
  2. Difference in water distribution (intra-/extracellular water, total water, overhydration) assessed by bioimpedance spectroscopy between patients with Primary Aldosteronism before treatment and healthy control subjects
Pulse wave velocity | 3 - 6 months after intervention
  1. Change in pulse wave velocity measured by SphygmoCor before and after treatment of Primary Aldosteronism
  2. Difference in pulse wave velocity between patients with Primary Aldosteronism before treatment and healthy control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kopp, MD, Principal Investigator — Nephrology Department, University Erlangen-Nurnberg, Germany
Locations (2):
- Germany (2):
  - Nephrology Department, University Hospital Erlangen, Erlangen, Bavaria
  - Radiology Department, University Hospital Erlangen, Erlangen, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kopp C, Linz P, Wachsmuth L, Dahlmann A, Horbach T, Schofl C, Renz W, Santoro D, Niendorf T, Muller DN, Neininger M, Cavallaro A, Eckardt KU, Schmieder RE, Luft FC, Uder M, Titze J. (23)Na magnetic resonance imaging of tissue sodium. Hypertension. 2012 Jan;59(1):167-72. doi: 10.1161/HYPERTENSIONAHA.111.183517. Epub 2011 Dec 5. PMID 22146510
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393